CLINICAL TRIAL: NCT03241303
Title: The Role of Glucagon-like Peptide-1 Receptor Signalling in the Glucose-lowering Effect of Increased Carbohydrate Content in the Distal Small Intestines After Meal Ingestion in Patients With Type 2 Diabetes
Brief Title: Delineation of the Role of Glucagon-like Peptide-1 Signalling in Relation to Increased Carbohydrate Content in the Distal Small Intestines
Acronym: AlfaEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Niels Bjørn Dalsgaard, Bachelor of Science, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-17007893
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Glucose Metabolism Disorders
Keywords: Glp-1; alpha-glucosidase inhibitor; acarbose
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — Acarbose; exendin (9-39)

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Acarbose (Experimental): 50 mg and 100 mg glucobay tablets. 2 weeks. Other name: Precose
  Interventions: Drug: Acarbose
- Placebo Oral tablets (Placebo Comparator): 180 mg. 2 weeks.
  Interventions: Drug: Placebo Oral Tablet
- Exendin (9-39) (Experimental): Infusion of GLP-1 receptor antagonist as a study tool to block GLP-1 activity on experimental day.
  Interventions: Drug: Exendin (9-39)
- Placbo Saline (Placebo Comparator): 9 mg/ml placebo saline infusion on experimental day.
  Interventions: Drug: Placebo Saline

INTERVENTIONS:
Drug: Acarbose — Glucobay tablets on experimental day.
  Other Names: Glucobay, Precose
  Arms: Acarbose
Drug: Placebo Oral Tablet — Placebo tablets on experimental day.
  Arms: Placebo Oral tablets
Drug: Exendin (9-39) — Infusion of GLP-1 receptor antagonist as a study tool to block GLP-1 activity on experimental day.
  Other Names: Ex(9-39)
  Arms: Exendin (9-39)
Drug: Placebo Saline — 9 mg/ml placebo saline infusion on experimental day.
  Arms: Placbo Saline

SUMMARY:
Investigation of GLP-1 signalling in the glucose-lowering effect of increased carbohydrate content in the distal small intestines induced by alpha-glucosidase inhibition during meal ingestion in patients with type 2 diabetes

DETAILED DESCRIPTION:
The primary aim of the study is to investigate whether GLP-1 released as a result of increased carbohydrate content in the distal and L cell-rich part of the small intestine after a meal affects postprandial plasma glucose levels in patients with type 2 diabetes. This will be done by applying an alpha-glucosidase inhibitor (to increase the postprandial carbohydrate content in the distal small intestine) and the specific GLP-1 receptor antagonist exendin(9-39) (to isolate any GLP-1-mediated effects) during meal tests in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least three months (diagnosed according to the criteria of the World Health Organization (WHO)) treated with metformin monotherapy
* Caucasian ethnicity
* Normal haemoglobin
* Age >18 years
* BMI >23 kg/m2 and <35 kg/m2
* Informed and written consent

Exclusion Criteria:

* Liver disease (alanine aminotransferase (ALAT) and/or serum aspartate aminotransferase (ASAT) >2 times normal values) or history of hepatobiliary disorder
* Gastrointestinal disease, previous intestinal resection, cholecystectomy or any major intra-abdominal surgery
* Reduced kidney function or nephropathy (estimated glomerular filtration rate (eGFR) <60 ml/min/1.73 m2 (based on serum creatinine) and/or albuminuria
* Treatment with medicine that cannot be paused for 12 hours
* Intake of antibiotics two months prior to study
* Treatment with glucose-lowering drugs other than metformin
* Hypo- and hyperthyroidism
* Treatment with oral anticoagulants
* Active or recent malignant disease
* Any treatment or condition requiring acute or sub-acute medical or surgical intervention
* Lack of effective birth control in premenopausal women
* Positive pregnancy test on study days in premenopausal women
* Pregnancy
* Women who are breastfeeding
* Any condition considered incompatible with participation by the investigators
* If the subjects receive any antibiotic treatment while included in the study they will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Plasma glucose | 240 min
  The primary outcome is the difference between the effect of increased carbohydrate content in the distal part of the small intestine (obtained by inhibiting alpha-glucosidase with acarbose) on postprandial glucose tolerance (as assessed by area under curve (AUC) for plasma glucose during a standardised liquid mixed meal test) with and without blockade of GLP-1 signalling by exendin(9-39).

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD, PhD, Study Director — University Hospital, Gentofte, Copenhagen
Locations (1):
- Center for Diabetesresearch, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No